CLINICAL TRIAL: NCT04328844
Title: First-in-Human Dose Study of IOA-244 in Patients With Advanced or Metastatic Cancers
Brief Title: A Study to Assess a PI3Kδ Inhibitor (IOA-244) in Patients With Metastatic Cancers
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: iOnctura (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IOA-244-101; 2019-000686-20 (EudraCT Number)
Record Dates: First submitted 2020-03-11; First posted 2020-03-31 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Solid Tumor, Adult; Non-Hodgkin Lymphoma, Adult; NSCLC; Myelofibrosis; Uveal Melanoma
Keywords: Mesothelioma; Melanoma; Follicular Lymphoma; NSCLC; Uveal Melanoma; Myelofibrosis; PTCL
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Primary Myelofibrosis; Uveal Melanoma; Mesothelioma; Melanoma; Lymphoma, Follicular | interventions — avelumab; Pemetrexed; Cisplatin; ruxolitinib

STUDY DESIGN:
Intervention Model Description: This is a two-part FIH dose study, where Part A is a dose-escalation group treatment study with IOA-244 and Part B is a parallel cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Group 1: Cutaneous Melanoma (Experimental): IOA-244 in combination with avelumab
  Interventions: Drug: IOA-244; Drug: Avelumab Injection
- Group 2: Uveal Melanoma (Experimental): IOA-244 as monotherapy
  Interventions: Drug: IOA-244
- Group 3: Myelofibrosis (Experimental): IOA-244 in combination with ruxolitinib
  Interventions: Drug: IOA-244; Drug: Ruxolitinib
- Group 4: Mesothelioma (Experimental): IOA-244 in combination with pemetrexed/cisplatin/avelumab
  Interventions: Drug: IOA-244; Drug: Avelumab Injection; Drug: Pemetrexed; Drug: Cisplatin
- Group 5: NSCLC 1st line (Experimental): IOA-244 in combination with pemetrexed/cisplatin/avelumab
  Interventions: Drug: IOA-244; Drug: Avelumab Injection; Drug: Pemetrexed; Drug: Cisplatin
- Group 6: NSCLC 2nd/3rd line (Experimental): IOA-244 in combination with avelumab
  Interventions: Drug: IOA-244; Drug: Avelumab Injection
- Group 7: NHL-FL and NHL-PTCL (Experimental): IOA-244 as monotherapy
  Interventions: Drug: IOA-244

INTERVENTIONS:
Drug: IOA-244 — IOA-244 will be administered orally once daily (QD)
Drug: Avelumab Injection — Avelumab will be administered IV every 2 weeks
  Arms: Group 1: Cutaneous Melanoma; Group 4: Mesothelioma; Group 5: NSCLC 1st line; Group 6: NSCLC 2nd/3rd line
Drug: Pemetrexed — Pemetrexed will be administered IV every 3 weeks
  Arms: Group 4: Mesothelioma; Group 5: NSCLC 1st line
Drug: Cisplatin — Cisplatin will be administered IV every 3 weeks
  Arms: Group 4: Mesothelioma; Group 5: NSCLC 1st line
Drug: Ruxolitinib — Ruxolitinib will be administered orally twice a day (BD)
  Arms: Group 3: Myelofibrosis

SUMMARY:
The objective of study IOA-244-101 is to determine whether IOA-244 is safe and tolerable in cancer patients (Part A). In addition, the study will assess whether IOA-244 can increase the anti-tumour immune response in patients both as monotherapy and in combination pemetrexed/cisplatin/avelumab (Part B Mesothelioma and NSCLC 1st line), in combination with avelumab (Part B Cutaneous Melanoma and NSCLC 2nd/3rd line) and ruxolitinib (Part B Primary Myelofibrosis)

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age inclusive, at the time of signing the informed consent.
2. Capable of giving signed informed consent, which includes compliance with the requirements of this protocol.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. For patients with NHL, ECOG 2 will be allowed.
4. Patients with histologically or cytologically confirmed advanced or metastatic malignancies (including histologically confirmed, unresectable Stage III or IV melanoma); see following details for each malignancy:

   For Patients with cutaneous and mucosal melanoma:
   1. Baseline lactate dehydrogenase levels are available.
   2. Disease progression is confirmed and they are eligible for second- or third-line treatment:

      * After first-line treatment and progression on approved programmed cell death-1 (PD-1) or cytotoxic T lymphocyte antigen-4 (CTLA-4) or combination of PD-1 and CTLA-4-pathway targeted agent.
      * After second-line treatment and progression on prior BRAF V600 mutation targeted agent followed by PD-1 or CTLA-4-pathway targeted agent (Note: There is no mandatory sequence of these approved treatments).
   3. No clinically significant tumour-related symptoms.

   For Patients with metastatic ocular/uveal melanoma:

   Patients must have metastatic histologically or cytologically confirmed uveal melanoma.

   For Patients with advanced or metastatic mesothelioma:
   1. Histological confirmation of mesothelioma (any subtype).
   2. Part A: They received at least one prior line of treatment (including patients who were re-challenged with pemetrexed-based therapy). Prior maintenance therapy is permitted but will not count as a line of treatment.

   Part B: Considered for first-line treatment with pemetrexed/cisplatin and avelumab.

   For Patients with Indolent Non-Hodgkin Lymphoma, type Follicular Lymphoma (FL):
   1. Patients must have a past diagnosis of indolent Non-Hodgkin lymphoma, type Follicular Lymphoma, Grade 1-3A.(Dreyling et al., 2016)
   2. Patients must have been previously treated with at least 1 prior systemic chemotherapy, immunotherapy, or chemoimmunotherapy, such as rituximab monotherapy, chemotherapy given with or without rituximab, radioimmunoconjugates (e.g., 90Y-ibritumomab tiuxetan and 131I-tositumomab).
   3. Must have documented relapsed, refractory, or PD after treatment with systemic therapy (refractory defined as less than PR or disease progression <6 months after last dose).
   4. Patients with prior exposure to a PI3K inhibitor (e.g., idelalisib/GS-1101, duvelisib) or a Bruton's tyrosine kinase (BTK) inhibitor are eligible if they discontinued either inhibitors in the last 4 weeks prior entering study treatment.
   5. Patients are not eligible for transplantation (autologous or any similar intervention, including CART-cell therapy).

   For Patients with Non-Hodgkin Lymphoma, type Peripheral T cell lymphoma (PTCL):
   1. Diagnosis of one of the following histologic subtypes of PTCL, pathologically-confirmed, as defined by the World Health Organization (other rare PTCL may be enrolled upon discussion with the medical monitor of this study):

      * Peripheral T-cell lymphoma - not otherwise specified (PTCL-NOS)
      * Angioimmunoblastic T-cell lymphomas (AITL)
      * Anaplastic large cell lymphoma (ALCL)
      * Natural-killer/T-cell lymphoma (NKTL)
   2. Received at least 2 cycles of one prior regimen administered with curative intent and one of the following:

      * failed to achieve at least a partial response after 2 or more cycles;
      * failed to achieve a complete response after 6 or more cycles; and/or
      * progressed after an initial response.
   3. For patients with CD30+ ALCL, failed or are ineligible or intolerant to brentuximab vedotin.
   4. Measurable disease as defined by IWG for PTCL, i.e., at least 1 measurable disease lesion > 1.5 cm in at least one dimension by 18FDG-PET-CT, MRI, or diagnostic CT.
   5. Patients with prior exposure to a PI3K inhibitor (e.g., idelalisib/GS-1101, duvelisib) or a Bruton's tyrosine kinase (BTK) inhibitor are eligible if they discontinued either inhibitors in the last 4 weeks prior entering study treatment.

   For Patients with Non-Small Cell Lung Cancer (NSCLC) 1st line:
   1. Histological diagnosis of locally advanced (primary or recurrent) NSCLC non-squamous not amenable for treatment with curative intent.
   2. No prior systemic treatment for unresectable locally advanced or metastatic disease for NSCLC.
   3. Non-squamous NSCLC, with no activating EGFR mutations, ALK or ROS1 translocations/rearrangements.
   4. If monotherapy pembrolizumab is available as a standard of care treatment option, patients must have a tumour proportion score (TPS) <50% for PD-L1 (e.g., via the 22C3 pharmDx or the Ventana (SP263) PD-L1 IHC assay, or any other approved IHC assay.

   For Patients with Non-Small Cell Lung Cancer (NSCLC) 2nd or 3rd line:
   1. Histological confirmed Stage IIIb/IV or recurrent NSCLC who have experienced disease progression.
   2. Considered for 2nd line or 3rd line treatment either after radiographic progression or on stable disease:

      * Participants must have progressed after a minimum of 2 cycles of 1 course of a platinum based combination therapy administered for the treatment of a metastatic disease.

   For Patients with Primary Myelofibrosis (PMF):
   1. Diagnosis of PMF, Post-Polycythemia Vera Myelofibrosis MF(PPV-MF), or post-essential thrombocythemia MF (PET-MF)
   2. Dynamic International Prognostic Scoring System (DIPSS) risk category of intermediate-1, intermediate-2, or high.
   3. Treated with ruxolitinib for ≥ 3 months with a stable dose for at least the last 8 weeks prior to Day 1 and no significant spleen reduction (e.g., less than 15% spleen size reduction, or corresponding lack of response in spleen volume).
   4. Did not receive experimental drug therapy for MF or any other drug considered as an effective treatment for MF (eg, danazol, hydroxyurea, interferon products) within the last 2 months prior to starting study treatment.
   5. Splenic irradiation within 6 months before receiving the first dose of study drug.
   6. Independent of spleen size. active symptoms of MF at the screening visit, as demonstrated by the presence of a Total Symptom Score (TSS) of ≥ 10 using the Screening Symptom Form.
   7. Screening bone marrow biopsy specimen and pathology report(s) available that was obtained no more than 2 months prior to starting the study treatment or willingness to undergo a bone marrow biopsy at screening/baseline; willingness to undergo bone marrow biopsy at Week 24 and every 24 weeks thereafter. Screening/baseline biopsy specimen must show diagnosis of MF.
   8. Peripheral blast count < 10%.
   9. Use of any potent CYP3A4 inhibitors or inducers within 14 days or 5 half-lives (whichever is longer) before the first dose of study drug or anticipated during the study.
5. Presence of measurable disease per RECIST v.1.1, or mRECIST (for cohort with pleural mesothelioma patients), as determined by the site study team. Tumour lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.

   For NHL (FL and PTCL) patients: Have measurable disease as defined by the Lugano Classification, including at least one lymph node or tumour mass greater than or equal to 1.5 cm.

   For PMF patients: Have measurable disease as defined by IWG-MRT criteria.
6. For patients with prior systemic therapies (Groups 1, 2, 6, and 7) disease progression must be reported after available therapies for advanced or metastatic disease that are known to confer clinical benefit, been intolerant to treatment, or refused standard treatment. Within 6 months and prior to entering the study, a patient who has completed an adjuvant, neo-adjuvant, or chemo-radiation regimens would be considered of having received 1 prior systemic regimen and would not require an additional systemic regimen for advanced or metastatic disease.
7. Willingness to undergo a pre-treatment and on-treatment tumour biopsy to obtain the specimen (for NHL and PMF: see respective requirements).

   Note: If a patient has signed the informed consent and is scheduled to have a tumour biopsy for the purposes of this study, and it is subsequently determined that tumour tissue cannot safely be obtained, the patient may still enrol in the study, and the patient may be replaced, if enrolled in Part A, after discussion between the Sponsor and Investigator. The patient will be replaced if enrolled in Part B. However, all patients will be part of the final safety PK, PD (except for the examinations related to the pre- and post-dosing biopsy) and efficacy evaluation.
8. Willingness to avoid pregnancy or fathering children based on the criteria below:

   1. Women of non-childbearing potential (i.e., surgically sterile with a hysterectomy and/or bilateral oophorectomy OR ≥ 12 months of amenorrhea and at least 50 years of age).
   2. Women of childbearing potential who had a negative serum pregnancy test at screening and who agree to take appropriate precautions to avoid pregnancy (with at least 99% certainty) from screening through safety follow-up, at least 1 month after the last dose of study treatment. Women receiving cisplatin should not become pregnant for at least 6 months after receiving the last dose of cisplatin. Permitted methods that are at least 99% effective in preventing pregnancy should be communicated to the patient and their understanding confirmed.
   3. Men who agree to take appropriate precautions to avoid fathering children (with at least 99% certainty) from screening through safety follow-up, at least 1 month after the last dose of study treatment. Men receiving pemetrexed and/or cisplatin should not father within 6 months of last treatment with pemetrexed and/or cisplatin. Permitted methods that are at least 99% effective in preventing pregnancy (see should be communicated to the patient and their understanding confirmed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2020-02-25 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Numbers of participants with treatment-related adverse events as assessed by CTCAE v5.0 | From time of first drug administration to first documented progression, toxicity or death from any cause whichever occurs first, assessed at week 30
  Adverse Events will be assessed by nondirective questioning of the participants during the screening process, at each visit during the study and during the safety follow up period

SECONDARY OUTCOMES:
Cmax | At Cycle 1 Day 1: 0 hours (pre-dose),1 hour, 2 hours, 3-4 hours and 6-8 hours post dose. From Cycle 2 Day 1 to Cycle 6 Day 1 (pre-dose). Each cycle is 28 days
  Peak Plasma Concentration
Cmin | At Cycle 1 Day 1: 0 hours (pre-dose),1 hour, 2 hours, 3-4 hours and 6-8 hours post dose. From Cycle 2 Day 1 to Cycle 6 Day 1 (pre-dose). Each cycle is 28 days
  Minimum observed plasma concentration
t½ | At Cycle 1 Day 1: 0 hours (pre-dose),1 hour, 2 hours, 3-4 hours and 6-8 hours post dose. From Cycle 2 Day 1 to Cycle 6 Day 1 (pre-dose). Each cycle is 28 days
  Terminal elimination half-life
tmax | At Cycle 1 Day 1: 0 hours (pre-dose),1 hour, 2 hours, 3-4 hours and 6-8 hours post dose. From Cycle 2 Day 1 to Cycle 6 Day 1 (pre-dose). Each cycle is 28 days
  Time of the maximum observed plasma concentration
AUC0-t | At Cycle 1 Day 1: 0 hours (pre-dose),1 hour, 2 hours, 3-4 hours and 6-8 hours post dose. From Cycle 2 Day 1 to Cycle 6 Day 1 (pre-dose). Each cycle is 28 days
  Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration
AUC0-∞ | At Cycle 1 Day 1: 0 hours (pre-dose),1 hour, 2 hours, 3-4 hours and 6-8 hours post dose. From Cycle 2 Day 1 to Cycle 6 Day 1 (pre-dose). Each cycle is 28 days
  Area under the plasma concentration-time curve from time zero extrapolated to infinity
Pharmacodynamic activity of IOA-244 by determining changes in Lymphocytes counts | At Cycle 1 Day 1, Day 2, Day 15 (pre-dose), From Cycle 2 to Cycle 6 Day 1 (pre-dose). Each cycle is 28 days
  Lymphocytes Immunophenotyping in peripheral blood
Pharmacodynamic activity of IOA-244 by determining changes in LDH | At Screening (D-28 to D-1), Cycle 1 Day 1, Day 8, Day 15, Day 22 (pre-dose). Each cycle is 28 days
  Levels of Lactate Dehydrogenase (LDH)
Pharmacodynamic activity of IOA-244 by evaluating levels of Mesothelin | At Cycle 1, Day 1 and Day 15 (pre-dose) , From Cycle 2 to Cycle 6, Day 1 (pre-dose). Each cycle is 28 days
  Levels of Mesothelin (Mesothelioma participants only)
Objective Response Rate (ORR) | Up to 28 weeks
  Percentage of participants with a Complete Response (CR) or Partial Response (PR) RECIST 1.1, for participants with Mesothelioma, modified RECIST and the Lugano 2014 criteria for NHL participants
Duration of response (DOR) | From date of the first documented evidence of CR or PR until the date of first documented disease progression or date of death from any cause, whichever came first, assessed up to 54 weeks
  DOR among patients who achieve objective response as determined by radiographic disease assessment
Progression Free Survival (PFS) | From date of the first dose of study treatment until the date of first documented disease progression or date of death from any cause, whichever came first, assessed up to 104 weeks
Overall Survival (OS) | From date of the first dose of study treatment until the date of death from any cause, assessed up to 150 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lahn, Study Director — iOnctura
Locations (3):
- Italy (2):
  - Humanitas Research Hospital, Rozzano, Milan
  - Medical Oncology and Immunotherapy Unit, University Hospital of Siena, Siena
- Beatson West of Scotland Cancer Centre, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No